CLINICAL TRIAL: NCT04063202
Title: A Longitudinal Study for Identifying Predictors of Incidence/Remission of Probable Depression and Developing a Predictive Index for Probable Depression Among Secondary School Students
Brief Title: Development of a Predictive Index for Probable Depression Among Secondary School Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HMRF16171001
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Depression; Stress; Youth
Keywords: Adolescent; Depression; Stress; Resilience
MeSH Terms: conditions — Depression | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-cases: Secondary school students (seventh to tenth years of education) without probable depression at baseline interview.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The anonymous structured questionnaire will be self-administered by the participating students in the absence of their teachers in class-room settings.

SUMMARY:
The present study aims to develop a new predictive index to predict future depression of adolescents by using factors including individual, interpersonal and environmental. The index can be used to predict likelihood of students who are non-probable depression cases convert into probable depression cases. In addition, the investigators also test the factors of depression remission. It can hence be used in school setting to identify high-risk students, and provide them with secondary interventions that are designed by considering modifiable significant variables identified in this unique, large-scale, longitudinal study.

DETAILED DESCRIPTION:
A 12-month longitudinal study will be conducted in secondary school settings.

The investigators will investigate incidence of probable depression (i.e., from non-depression, CESD<16, at baseline to probable depression, CESD≥16, at month 12) and remission of probable depression.

The investigators will investigate factors that can prospectively predict new cases/remission of probable depression, including both well-documented risk/protective factors and some under-examined but potentially important local factors (e.g. school/academic stress, psychological resilience). The relative importance of the risk/protective factors at different socio-ecological levels will be compared and their combined effect will be identified.

Based on the selected factors, the investigators will derive a new prediction index called the Adolescent Depression Prediction Index (ADPI) in a model building sample and test its performance in predicting incidence of depression in a validation sample among secondary school students in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Secondary 1 (seventh year of formal education) to Secondary 4 Chinese students, who are studying local mainstream schools in Hong Kong.
* Able to read Chinese and speak either Cantonese or Mandarin.

Exclusion Criteria:

* Eligible students whose parents refuse to give consent to take part in the study.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Out of the 18 districts in Hong Kong, nine randomly selected districts will select randomly two schools and while the rest nine will randomly select one school. Replacements of schools will be made upon refusals. Within the selected schools, all Secondary 1-4 students will be invited to join the study. Students will be asked to fill in baseline questionnaires in the absence of teachers in classroom settings.
Sampling Method: Probability Sample
Enrollment: 4799 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of probable depression | 12 months
  To examine the incidence of probable depression from non-depression (CESD<16) at baseline to probable depression (CESD>=16) at month 12.
Adolescent Depression Prediction Index (ADPI) | 12 months
  To develop a new prediction index ADPI and test test its performance in predicting incidence of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yang, PhD, Principal Investigator — JC School of Public Health and Primary Care, Faculty of Medicine, CUHK
Locations (4):
- Hong Kong (4):
  - China Holiness Church Living Spirit College, Hong Kong
  - Christian Alliance SW Chan Memorial College (Christian Alliance SW Chan Memorial Secondary School), Hong Kong
  - Ho Ngai College ( Sponsored By Sik Sik Yuen), Hong Kong
  - Kit Sam Lam Bing Yim Secondary Schoo, Hong Kong

IPD SHARING:
Plan to Share IPD: No